CLINICAL TRIAL: NCT04820608
Title: Epithelium-on Customized Cross-linking for Keratoconus
Brief Title: Transepithelial Customized Cross-linking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ophthalmica Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OphthalmicaEI
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Keratoconus
Keywords: keratoconus; cross-linking; transepithelial; oxygen-boosted; customized; CXL
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Customized, transepithelial cross-linking (Experimental): All study patients will be treated according to the customized remodeled vision protocol
  Interventions: Device: Cross-linking

INTERVENTIONS:
Device: Cross-linking — Oxygen-boosted, epithelium-on, customized cross-linking. Highest UV-A application is focused on the apex of the cone. The cone area receives a moderate amount of UV-A, while healthy cornea is spared.
  Other Names: Customized remodeled vision

SUMMARY:
Customized remodeled vision (CuRV) is a new corneal cross-linking protocol for keratoconus, combining a transepithelial approach with customized energy application. Our aim is to follow-up our patients and establish the short-and long-term results of CuRV.

DETAILED DESCRIPTION:
Customized remodeled vision is a protocol for oxygen-boosted, tranespithelial cross-linking, customized to apply higher energy at the apex of the cone, relatively lower to the cone area and none to healthy cornea. Thus CuRV promises to halt keratoconus progression, simultaneously offering potential for relatively good visual rehabilitation.Our primary outcomes involve spectacle-corrected distance visual acuity and changes in corneal topography/tomography and OCT parameters. These parameters include Kmax, thinnest corneal pachymetry, maximal anterior and posterior elevation, the Fourier analysis-derived irregularity index, and demarcation line depth.

ELIGIBILITY:
Inclusion Criteria:

* Topographic evidence of keratoconus:
* maximum corneal curvature (Kmax) ≥47.00 D,
* localized steepening on topographic maps,
* localized elevation in the anterior and posterior corneal surfaces.

Exclusion Criteria:

* Hypersensitivity to riboflavin
* Thinnest corneal pachymetry < 380 μm
* History of corneal surgery, including previous cross-linking
* Corneal scarring
* Aphakia
* Pseudophakia
* Any visually significant ocular condition

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Spectacle-corrected distance visual acuity | 1-3-6 months, 1 year, 2 years
  Measurements will be performed on Early Treatment of Diabetic Retinopathy Study charts in logMAR units
Kmax | 1-3-6 months, 1 year, 2 years
  Maximal corneal keratometric value measured on Scheimpflung corneal tomography

SECONDARY OUTCOMES:
Demarcation line depth | 1 month
  Measurements will be performed at 1st postoperative month, when the demarcation line is most visible, on anterior segment optical coherence tomography. The measurement will be performed manually on the scan approximating the thinnest corneal location with the device-native caliper set at 1:1μm.
Thinnest corneal pachymetry | 1-3-6 months, 1 year, 2 years
  Values as indicated on Scheimpflung corneal tomography device
Maximal anterior & posterior elevation | 1-3-6 months, 1 year, 2 years
  Values as indicated on the Belin Ambrosio Enhanced Ectasia module of the Scheimpflung tomography device
Fourier analysis-calculated maximum decentration | 1-3-6 months, 1 year, 2 years
  Values as indicated on the Fourier analysis module of the Scheimpflung tomography device
Regularization index | 1-3-6 months, 1 year, 2 years
  Regularization index was proposed by Seiler et al. The measurement will be performed using the maximum flattening and steepening on the Comparison display of the Scheimpflung tomography device.

CONTACTS AND LOCATIONS:
Overall Officials: Miltos Balidis, PhD, Principal Investigator — Ophthalmica Eye Institute
Locations (1):
- Ophthalmica Eye Institute, Thessaloniki, Kalamaria, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seiler TG, Fischinger I, Koller T, Zapp D, Frueh BE, Seiler T. Customized Corneal Cross-linking: One-Year Results. Am J Ophthalmol. 2016 Jun;166:14-21. doi: 10.1016/j.ajo.2016.02.029. Epub 2016 Mar 2. PMID 26944278